CLINICAL TRIAL: NCT05066581
Title: Vitoria Sleep Smart City: Interactive Intervention for Sleep Improvement.
Acronym: SMARTCITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Araba (Other)
Collaborators: Philips Healthcare (Industry); Ayuntamiento de Vitoria (Unknown); Ibermatica (Unknown); Bioaraba (Unknown)
Responsible Party: Principal Investigator, Carlos Javier Egea Santaolalla,Ph, HEAD OF FUNCTIONAL SLEEP UNIT, Hospital Universitario Araba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: PI21/0108
Record Dates: First submitted 2021-09-08; First posted 2021-10-04 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Sleep Deprivation; Sleep Hygiene
MeSH Terms: conditions — Sleep Deprivation; Sleep Hygiene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Philips band (No Intervention): It is a medical device that collects, among other things, movement data by means of an accelerometer, from which it accelerometer, from which it estimates the total time of sleep (TTS) and wakefulness, and waking time, also offering the efficiency of the same (time asleep in relation to time in bed). time in bed). In addition, it collects data not related to sleep, such as energy expenditure (in kilocalories), energy expenditure (in kilocalories) (in kilocalories), heart rate, and daily activity (in steps), among others.
- Philips Band + Live chat (Active Comparator): In the Intervention group, in addition to having the philips band, the subjects will interact through the live chat system that they will have to download to their mobile phones. This live chat offers the possibility to consult in real time, thus initiating a process of relationship between researcher/subject.
  Interventions: Device: Live Chat

INTERVENTIONS:
Device: Live Chat — Subjects from the intervention group will be able to ask for a medical intervention if needed with the phisycians from the sleep unit. After the following period, we expect to see better sleep habits in this group when compared to the no intervention one
  Arms: Philips Band + Live chat

SUMMARY:
Currently, the investigators know that there is a high and increasing prevalence of sleep quality and quantity deficits in the general population with the social and health consequences that this entails. There are numerous activity wristbands linked to mobile apps that analyze sleep, but none can generate individualized recommendations for improvement interacting with the person. The main objective of the current project is to develop a virtual and interactive sleep assistant to increase the quantity and quality of sleep. Secondary objectives being the improvement of daytime sleepiness and the quality of life of the persons.

Methodology: 202 participants in active employment who meet the criteria of "poor sleepers" (defined by a Pittsburg test score >5) are divided into 2 study groups. 1. Intervention group: Sleep data will be collected using validated questionnaires (SATED and the Sleep Hygiene Index) and objectively employing an activity bracelet, in which weekly, through a live chat, the medical staff of the sleep units will offer recommendations for the improvement of the deficits detected. 2. Control group: Same protocol as the intervention group, but the participants will not receive the recommendations via the interactive chat.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65 years

Exclusion Criteria:

* Patients previously diagnosed and treated for sleep pathology (such as insomnia, Obstructive Sleep Apnea (OSA), Restless Legs Syndrome (RLS), narcolepsy or parasomnia, among others).
* Severe medical or psychiatric comorbidities.
* Subjects who are not capable of using mobile technology such as Smartphone.
* Subjects who are not committed to actively participate, putting into practice the sleep recommendations given by the assistant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Total sleep time | Eight months
  By measuring total sleep time, determine the objective of sleeping between 7 and 9 hours per day on average.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Alava, Vitoria-Gasteiz, Alava, Spain

IPD SHARING:
Plan to Share IPD: No